CLINICAL TRIAL: NCT02319460
Title: An Observational Cohort Study of the Risk of Thromboembolic Events Among Adult Patients Treated With KCENTRA® Compared With Plasma for Urgent Reversal of Vitamin K Antagonist Therapy in the Setting of Acute Major Bleeding
Brief Title: An Observational Cohort Study to Investigate the Risk of Thromboembolic Events in Patients Receiving Kcentra® or Plasma to Reverse Vitamin K Antagonist (VKA) Therapy in the Setting of Acute Major Bleeding
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: BE1116_4001
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Hemorrhage
Keywords: Vitamin K Reversal Antagonist Therapy of Acute Major Bleeding; Warfarin Reversal
MeSH Terms: conditions — Hemorrhage | interventions — Factor IX; factor IX, factor VII, factor X, prothrombin drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Retrospective: Retrospective cohort of adults hospitalized for major bleeding during 2008 to 2013 who receive plasma for urgent reversal of acquired coagulation factor deficiency induced by oral VKA therapy
  Interventions: Biological: Plasma
- Prospective: Prospective parallel cohort of adults hospitalized for major bleeding during 2014 to 2020 who either receive Kcentra® or plasma for urgent reversal of acquired coagulation factor deficiency induced by oral VKA therapy
  Interventions: Biological: Kcentra®; Biological: Plasma

INTERVENTIONS:
Biological: Kcentra® — Kcentra®, Prothrombin Complex Concentrate (Human), is a blood coagulation factor replacement product that contains coagulation Factors II, VII, IX and X, and antithrombotic Proteins C and S as a lyophilized concentrate.
  Other Names: Prothrombin Complex Concentrate (Human); Beriplex
  Groups: Prospective
Biological: Plasma

SUMMARY:
This observational cohort study is designed to obtain product safety information from the routine clinical setting within large, diverse, community-based populations. In the setting of acute major bleeding in which patients are treated for Vitamin K antagonist reversal, the risk of thromboembolic events (TEE) in patients treated with Kcentra® and in patients treated with plasma will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older at admission for VKA-associated major bleeding
* A minimum of 365 days of continuous health plan enrollment before the index hospitalization involving acute VKA reversal treatment
* A minimum of 365 days of continuous pharmacy benefit before the index hospitalization involving acute VKA reversal treatment

Exclusion Criteria:

Patients will be excluded from the primary analyses if they:

* Require urgent reversal of VKA therapy in the setting of bleeding due to major trauma (eg, motor vehicle accident)
* Requiring urgent reversal of VKA therapy for a surgical procedure unrelated to major bleeding (eg, appendicitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult members of the Kaiser Permanente Northern and Southern California health care delivery systems, receiving chronic warfarin therapy and meeting study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2238 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Risk of thromboembolic events (TEE) for patients without a recent history of TEE | Within 45 days after the index date
  The risk of confirmed thromboembolic events (TEE) will be estimated for patients without a recent history of TEE treated with Kcentra® compared to patients treated with plasma. The index date is the date of acute VKA reversal for major bleeding event.

SECONDARY OUTCOMES:
Risk of thromboembolic events | Within 45 days after the index date
  The risk of confirmed TEE and confirmed fatal TEE will be each estimated for patients treated with Kcentra® compared to patients treated with plasma, overall and for patients in the following subgroups:
  * Recent history of TEE
  * No recent history of TEE
  * Any history of TEE
  The index date is the date of acute VKA reversal for major bleeding event.
Risk of death from any cause | Within 45 days after the index date
  The risk of death from any cause will be estimated for patients treated with Kcentra® compared to patients treated with plasma, overall and for patients in the following subgroups:
  * Recent history of TEE
  * No recent history of TEE
  * Any history of TEE
  The index date is the date of acute VKA reversal for major bleeding event.
Rates of use of VKA therapy after the index date | Within 90 days after the index date
  The rates of use of VKA therapy or other antithrombotic agents will be assessed among patients with and without any history of TEE. The index date is the date of acute VKA reversal for major bleeding event.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Epidemiologist, Study Director — CSL Behring; Alan S. Go, MD, Principal Investigator — Kaiser Permanente; Kristi Reynolds, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Study Site, Oakland, California, United States